CLINICAL TRIAL: NCT04808232
Title: The Effect of Health Education and Progressive Muscle Relaxation Exercise on Vasomotor Symptoms and Sleep Problems in Women With Perimenopausal Period
Brief Title: The Effect of Health Education and Progressive Muscle Relaxation Exercise on Vasomotor Symptoms and Sleep Problems With Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidika Pelit Aksu (Other)
Responsible Party: Sponsor-Investigator, Sidika Pelit Aksu, Research asistant (RN), Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 168846
Record Dates: First submitted 2021-03-13; First posted 2021-03-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Vasomotor Symptoms; Hot Flashes; Sleep Problem
Keywords: Vasomotor symptoms,; sleep problems,; health education,; progressive muscle relaxation exercise
MeSH Terms: conditions — Hot Flashes; Parasomnias; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- health education and progressive muscle relaxation exercise (Experimental): Health education and progressive muscle relaxation exercise training was given to women in this group.
  Interventions: Behavioral: progressive muscle relaxation exercise
- progressive muscle relaxation exercise (Experimental): Progressive muscle relaxation exercise training was given to women in this group.
  Interventions: Behavioral: progressive muscle relaxation exercise
- Control group (No Intervention): women in this group were not intervened.

INTERVENTIONS:
Behavioral: progressive muscle relaxation exercise — We used "the muscle relaxation audio CD" produced by the Turkish Psychologists Association. The CD consists of three parts; the 10-min first part includes definition and purpose of relaxation, and points to take into consideration during relaxation, the 30-min second part includes instructions with river sounds, and the 30-min third part includes only relaxing music without instructions. We used the second part of the audio record in this study. Following the instructions on the CD, the students tensed each muscle group from hands to feet, and then, all muscles in their face and body for approximately 10 s. The women breathed in, tensed a specific muscle group, and then relaxed it while breathing out. The relaxation step took 10-20 s before tensing the next muscle group. Thus, the women relaxed by tensing and relaxing the muscle groups in hands, arms, neck, shoulder, chest, stomach, hips, foot and fingers, and all muscles in the face and body.
  Other Names: health education
  Arms: health education and progressive muscle relaxation exercise; progressive muscle relaxation exercise

SUMMARY:
This study aims to determine the effect of health education and progressive muscle relaxation exercise (PMRE) on vasomotor symptoms and sleep problems in women with perimenopausal period; a randomized, pretest-posttest is a randomized controlled, factorial group experimental study. The research was conducted in a family health center. The required institutional permission and ethics committee approval was received. The sample consisted of 90 women totally, 30 of whom in the PMRE + health education group, 30 of whom in the PMRE group and 30 of whom in the control group. The data was collected using personal information form, Visual Analog Scale for Vasomotor Symptoms (VAS), Women's Health Initiative Insomnia Rating Scale-WHIIRS, vasomotor symptom diary, progressive muscle relaxation exercise follow-up schedule, and health education practice follow-up schedule. The data were stored in the SPSS 24 program. In the analysis of the data, ANOVA test, Repeated Measures test, Kruskal-Wallis H test, Friedman test and χ2 test statistics were used.

DETAILED DESCRIPTION:
Purpose and type of study The study examines the effects of health education and progressive muscle relaxation exercise (PMRE) on vasomotor symptoms and sleep problems in women in the perimenopausal period; pretest-posttest is a randomized controlled, factorial group experimental study.

Universe and sample The research was conducted in a family health center. The required institutional permission and ethics committee approval was received. The universe of the research consists of 1830 women between the ages of 40-55 registered at Gazi Family Health Center. A pilot application was conducted to determine the sample size in the study. Power analysis was performed using the G * Power 3.0.10 program with 18 women (PMRE + Health education group (n = 6), PKGE group (n = 6), control group (n = 6)) who took part in the pilot study. According to the power analysis performed by calculating the effect size (0.177), the sample size calculated with 90% power and 5% margin of error; A total of at least 84 women were identified, including 28 women in the PMRE + Health education group, 28 women in the PMRE group and 28 women in the control group. Similar to our study, 36 women were included in each group in our study by calculating the drop-out rate in the study of Garcia et al. (2018) (Garcia et al., 2018).

The data collection process of the research started on 17.02.2019 and the determined sample number was completed on 02.04.2020. In this process, women who applied to ASM between 17.02.2019-23.01.2020 and who met the sampling criteria and accepted to participate in the study after the purpose and importance of the study were explained were determined. Under the direction of the researcher, the women interviewed a nurse independent of the study. Nurse The inclusion criteria used the check-list form to evaluate the compliance of the women with the research criteria. Personal information form, vasomotor symptom VAS and Women's Health Initiative Insomnia Scale-WHIIRS (pre-tests) were applied to determine compliance with the criteria. After the women meeting the criteria were informed about the study and consent was obtained, randomization was performed. During the study, a total of 482 women who applied to family health center were interviewed. Of these women; non-perimenopausal (n = 20), surgical menopause (n = 17), using psychiatric drugs and sleeping pills (n = 62), using alcohol (n = 14), women health initiative insomnia scale score below 10 (n = 78), the severity score of VAS symptoms for vasomotor symptoms is less than 3 (n = 69), who received hormone replacement therapy (n = 27), the number of moderate and severe hot flashes per day (n = 67), and A total of 374 women who did not agree to participate in the study (n = 20) were not included in the study. A total of 108 women who met the research criteria were stratified according to their smoking and regular exercise status. After stratification, women were assigned to the groups by simple randomization method (closed envelope method). For this purpose, three different envelopes were formed by placing the cards with A, B and C in the envelopes. A: PMRE + Health education group, B: PMRE group, C: represent the control group. In order to prevent bias and hide randomization, random assignments were made to the groups by the nurses using the closed envelope method. According to the envelope result, women were included in the PMRE + Health education group, the PMRE group and the control group. The study sample included women in the PMRE + Health education group (n = 36), the PMRE group (n = 36), and the control group (n = 36). Women participated in the practices prepared for the groups they were included in. Six of the women in the PMRE + Health education group participated in the training, but were excluded from the sample due to moving (n = 2), death of a relative (n = 1), illness (n = 1) and not doing PMRE in sufficient numbers (n = 2). Six of the women in the PKGE group participated in the training, but were excluded from the sample due to the death of the relative (n = 1) and the illness (n = 2) not making PKGE sufficiently (n = 3). Six women in the control group were excluded from the sample because they would voluntarily (n = 4) and start a new job (n = 2). As a result; A total of 18 women included in the sample left the study, the study was completed with women in the PKGE + Health education group (n = 30), the PMRE group (n = 30), and the control group (n = 30). At the end of the research; As a result of the power analysis made using the G * Power 3.0.10 program; At least 90 women in total were found to be sufficient with 90% power, 5% margin of error and 0.172 effect size.The data was collected using personal information form, Visual Analogue Scale for Vasomotor Symptoms (VAS), Women's Health Initiative Insomnia Rating Scale-WHIIRS, vasomotor symptom diary, progressive muscle relaxation exercise follow-up schedule, and health education practice follow-up schedule.

Randomization In our study, support was received from a statistician during the randomization phase. The stratified sampling method was applied over these two prognostic factors to ensure randomization, as it is thought that smoking (smoker and non-smoker) and regular exercise (regularly exercising and not exercising regularly) may affect our study results. After stratification; A total of four groups were determined according to the layer properties.

Four stratum groups were formed to ensure equal distribution of women in terms of smoking and regular exercise in the experimental and control groups in the study. The closed-envelope method was used to assign stratified women to the control and experimental groups without being biased, and an equal number of women were assigned to each group. During the preparation of envelopes, opaque envelopes are used to prevent the inside of the envelope from being seen from the outside. The envelopes were created by a nurse working at the Family health center, independent of the research. Three different envelopes were formed by placing the cards A, B and C in the envelopes. A: PMRE + Health education group, B: PMRE group, C: represents the control group. In order to prevent bias and conceal randomization, women were randomly assigned to the groups by a sealed envelope method by a second nurse working at family health center outside the researcher. The nurse placed women who met the research criteria in the appropriate strata from four strata. When groups of three people were formed in each stratum, the women from the strata were assigned to the groups as follows. He asked the first woman with the same characteristics to come to each stratum group to pull one of the three envelopes marked A, B, and C. For example: If C is in the envelope, the first woman who came was assigned to the control group. For the second woman, she was asked to pull one of the two envelopes, this time marked A and B. If A was placed in the draw, the second woman was assigned to the PMRE + Health education group. The envelope was not drawn for the third woman who came, and she was assigned to the last remaining group, the PMRE group. The same method was applied for all three women in the same layer after that.

Thus, 108 women in the sample were randomly assigned to the PMRE + Health education group, the PMRE group and the control groups stratified and equally. Until the initiatives started, the groups to which the women were assigned were not known to the researchers. The homogeneity of the randomized groups was compared with the chi-square test and it was found that there was no statistical difference between the groups in terms of stratification criteria, and the groups were homogeneous.

Prevention of bias In the study, women in the PMRE + Health education group and the PMRE group could not be blinded because they will participate in the training. In order to prevent bias, women were informed, assigned to groups and data were collected by a nurse outside of the study. However, the study was carried out by the researcher because the research was a thesis study, the number of application groups was high, multiple attempts were applied and the application should be done by an experienced researcher. For these reasons, the researcher could not be blinded. Prevention of bias in the research (in terms of data collectors, statistician and reporting) has been done. The pre and post-tests were filled by a nurse independent of the research. The collected data were coded as A, B and C groups by the researcher in a package program called SPSS (IBM SPSS Statistics 24). The analysis of the data coded in terms of groups was done and reported by a statistician. In this way, detection bias, statistical bias, and reporting bias were controlled.

Data collection and application process

1. st evaluation (conducted in the 1st week) The women who applied to the family health center and met the sampling criteria and accepted to participate in the study after the purpose and importance of the study were explained were determined. The women were informed about the research by the nurse with the direction of the researcher. Nurse 'The inclusion criteria used the check-list form to evaluate the compliance of the women with the research criteria. It was ensured that women filled the personal information form, vasomotor symptom VAS and Women's Health Initiative Insomnia Scale, which are necessary to determine compliance with the criteria. The nurse placed the women who met the criteria in the appropriate strata from four strata. When groups of three people were formed in each stratum, women were assigned to the groups as follows. He asked the first woman with the same characteristics to come to each stratum group to pull one of the three envelopes marked A, B, and C. For example; If C is in the envelope, the first woman arriving was assigned to the control group. For the second woman, she was asked to pull one of the two envelopes, this time marked A and B. If A was placed in the draw, the second woman was assigned to the PMRE + Health education group. The envelope was not drawn for the third woman who came, and she was assigned to the last remaining group, the PMRE group. The same method was applied for all three women in the same layer after that. Thus, women were randomly assigned to the study groups.

   Following this, a vasomotor symptom diary was given to all women by the nurse. The women assigned to the PMRE + health education group and the PMRE group were asked to complete the vasomotor symptom diary every day for a week until a training class would be established one week later and up to this training class. The women in the control group were instructed to fill in the vasomotor symptom diary until the end of the study. The averages in the diary filled in the first week of all women formed the baseline data before starting the study.

   Establishment of PMRE + health education and PMRE education classes (1st week was held) When small groups of 3 people are formed in the stratification groups and 3 women are appointed to the working groups, by taking name lists from the nurse; The researcher interviewed women. In these meetings; An explanation and planning were made for the groups to be intervened about the training day, place, time, duration, and wearing appropriate/comfortable clothes. At the beginning of the second week of the study, a time frame between 13.00-16.00 was determined to be suitable for the researcher and all three women in his group. In PMRE + Health education and PMRE group, training was given in groups of three (12 groups + 12 groups = 24 groups). The application was made in a room allocated for research in the family health center. This room is quiet, dim, and spacious. There are seats and a table for women and the researcher. Considering the capacity of this room, it was decided that it would be appropriate for the groups to have three people in order for women to participate in health education more actively and the researcher could observe each woman performing PMRE in detail. The women were asked to attend the training in comfortable clothes and not to be very hungry or full. The hall is pre-ventilated for the application and the application environment has been prepared. In order not to be disturbed during the application, a warning letter is hung on the door. Participants were offered water during the training sessions, tea, chocolate, sweets, dried fruits, cakes, etc. after the application.

   Training the PMRE + health education group (2nd week) Each group was provided with health education (training on vasomotor symptoms and sleep hygiene) and PMRE practice training. Health education (training on vasomotor symptoms and sleep hygiene) lasted approximately 30 minutes. Then, the gradual muscle relaxation exercise was performed by the researcher in line with the musical instruction prepared by the Turkish Psychologists Association (01.01.2010) for 30 minutes. After an interval of approximately 10 minutes, PMRE was performed by women for approximately 30 minutes.

   The training started with health education (training on vasomotor symptoms and sleep hygiene). The researcher will spend about 30 minutes with a slide show prepared in accordance with the content of the educational guide. He gave training. During and after the training, questions from women were answered, women's own experiences were shared, and they were talked about how to apply education to their daily lives. The questions of women who were hesitant about this issue or who thought they might have trouble at the point of the application were answered. Participants in the training were given a booklet titled "A Guide to Coping with Hot Flashes, Night Sweats, and Sleep Problems Frequently Encountered in the Transition to Menopausal Period" prepared by the researchers. At the end of the training, the women were asked to apply the topics of health education to their daily lives as much as possible every day for 8 weeks, if not at least 4 days a week. It was stated that those who do not comply with this program will be excluded from the sample.

   The researcher first demonstrated the PMRE application by doing it himself and then enabled the participants to practice. All participants were observed by the researcher during the learning process and they were ensured to apply progressive muscle relaxation exercises correctly. At the end of the exercise, the women were asked to do relaxation exercises every day if possible for 8 weeks, at least 4 times a week when this was not possible, before going to sleep at night. The musical instructions for the gradual relaxation exercise were uploaded to the phones of all women. Feedback was obtained from the women after the first exercise alone and the questions were answered. Thus, women were provided to do the application correctly.

   A Whatsapp® group was established for each 3-person training group in order to monitor and encourage women to exercise health education and exercise. The women were asked to report from this group when they adapted their health education to their daily lives and after applying the exercise. Throughout the study, the women were reminded to adapt health education and exercise every day from the Whatsapp® group, and women who did/did not practice the application were identified with their feedback.

   At the end of the training given by the researcher, the women were given a vasomotor symptom diary, PMRE follow-up chart, and health education follow-up chart to fill in until the end of the study. Women marked their practices on the health education follow-up chart and progressive muscle relaxation exercise follow-up chart for 8 weeks. This marked chart was retrieved from the participants at the end of the 8-week practice.
2. nd evaluation (made in the 5th week) Four weeks after the PMRE + health education, women were made to fill the Women's Health Initiative Insomnia Scale and the visual analog scale for vasomotor symptoms for the second time by the nurse. They were reminded to continue filling out the diary and charts until the research was completed.
3. rd evaluation (conducted at the 9th week)

8 weeks after the PMRE + health education, the nurse was asked to fill the Women's Health Initiative Insomnia Scale and the visual analog scale for vasomotor symptoms for the third and last time. The diaries and charts they filled out were taken and filed, and the research was terminated. The data were collected as specified in the application calendar.

Training the PMRE group (2nd week) Only women in the PMRE group were taught how to perform PMRE. Approximately 30 minutes, the gradual muscle relaxation exercise was applied by the researcher in accordance with the musical instruction prepared by the Turkish Psychological Association (01.01.2010). Then, women were allowed to apply PMRE for approximately 30 minutes.

All participants were observed by the researcher during the learning process and they were ensured to apply progressive muscle relaxation exercises correctly. At the end of the exercise, the women were asked to do relaxation exercises every day if possible for 8 weeks, at least 4 times a week when this was not possible, before going to sleep at night. The musical instructions for the gradual relaxation exercise were uploaded to the phones of all women. Feedback was obtained from the women after the first exercise alone and the questions were answered. Thus, women were provided to do the application correctly.

In order to monitor and encourage women to do PMRE, a Whatsapp® group was established for each 3-person training group. The women were asked to report from this group after applying the exercise. Throughout the study, women were reminded to do the exercise every day, and women who did/did not do it were identified with their feedback.

At the end of the training given by the researcher, the women were given a vasomotor symptom diary and PCI follow-up chart to fill in until the end of the study. Women marked their practices on the Progressive Muscle Relaxation Exercise Follow-up Chart for 8 weeks. This marked chart was retrieved from the participants at the end of the 8-week practice.

2nd evaluation (conducted at the 5th week) Four weeks after the training, women were made to fill the Women's Health Initiative Insomnia Scale and the visual analog scale for vasomotor syndromes for the second time by the nurse at the Family health center. They were reminded to continue filling out the diary and charts until the research was completed.

3rd evaluation (conducted at the 9th week) 8 weeks after the training, women were provided to fill the Women's Health Initiative Insomnia Scale and the visual analog scale for vasomotor symptoms for the third and last time by the nurse at the family health center. The research was concluded by taking the diary and charts they filled out. The data were collected as specified in the application calendar.

Control group

1. st evaluation (conducted in the 1st week) In the first evaluation, women were made to fill in the personal information form, vasomotor symptom VAS, and the Women's Health Initiative Insomnia Scale. After the pre-tests were applied, random assignments were made to the groups. Following this, a vasomotor symptom diary was given to women in the control group by the nurse. They were instructed to fill in the vasomotor symptom diary until the end of the study. No intervention was applied to the women assigned to the control group as a result of randomization.
2. nd evaluation (conducted at the 5th week) The nurse made it possible for women to fill the Women's Health Initiative Insomnia Scale for the second time and the visual analog scale for vasomotor symptoms. They were reminded to continue filling in the diary until the end of the study.
3. rd evaluation (conducted at the 9th week) women were provided to fill the Women's Health Initiative Insomnia Scale and the visual analog scale for vasomotor symptoms for the third and last time by the nurse. The research was terminated by taking the diaries they filled. The data were collected in accordance with the application schedule.

The data were stored in the SPSS 24 program. In the analysis of the data, ANOVA test, Repeated Measures test, Kruskal-Wallis H test, Friedman test, and χ2 test statistics were used.

ELIGIBILITY:
Inclusion Criteria:

* Being in the perimenopausal period according to the Staging of Reproductive Aging in Women (STRAW) criteria,

  * Women in the early menopause transition phase (STRAW -2). In these women, there is a variation in the duration of the cycles for 7 days or more.
  * Women in the late menopausal transition phase (STRAW -1). These women have amenorrhea that lasts 60 days or longer.
* Having entered natural menopause,
* Not receiving hormone replacement therapy in the past and / or currently,
* Not having a diagnosed psychiatric disease,
* Not using alcohol,
* Not using sleeping pills,
* Not doing any other body-mind based practice (meditation, hypnosis, yoga, mindfulness techniques-minfulness, guided imagery technique), Not having a disease that may cause sleep problems and vasomotor symptoms and not receiving medical treatment (thyroid diseases, heart failure, neurological disorders),
* Women health initiative insomnia scale score above 10,
* VAS severity score above 3 for vasomotor synptomes,
* Number of moderate and severe hot flashes over 3 a day,
* To have a smart mobile phone (IOS and Android) and to be using it effectively

Exclusion Criteria:

* Failure to communicate by calling 3 times on different days during the follow-up and the woman not returning to the phone call
* Woman not applying PMRE and health education at most 3 times a week
* The woman leaves the research voluntarily.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
daily night sweats frequency | 9 weeks
  daily night sweats frequency
daily hot flashes frequency | 9 weeks
  daily hot flashes frequency
mean VAS score for hot flashes and night sweats | 9 weeks
  mean VAS score for hot flashes and night sweats
the mean sweating VAS score | 9 weeks
  the mean sweating VAS score
mean daily hot flash and night sweats severity score | 9 weeks
  mean daily hot flash and night sweats severity score
Women's Health Initiative Insomnia Scale mean score | 9 weeks
  Women's Health Initiative Insomnia Scale mean score

CONTACTS AND LOCATIONS:
Locations (1):
- Sıdıka PELİT AKSU, Ankara, Turkey/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelit Aksu S, Senturk Erenel A. Effects of health education and progressive muscle relaxation on vasomotor symptoms and insomnia in perimenopausal women: A randomized controlled trial. Patient Educ Couns. 2022 Nov;105(11):3279-3286. doi: 10.1016/j.pec.2022.07.015. Epub 2022 Jul 28. PMID 35961801